CLINICAL TRIAL: NCT01148290
Title: A Comparison Between Tension-free Vaginal Tape and Bulking Agent for the Treatment of Post-vulvectomy Urinary Incontinence: a Randomized Controlled Trial
Brief Title: Tension-free Vaginal Tape (TVT) Versus Bulking Agent for the Treatment of Post Vulvectomy Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03/2010
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Urinary Incontinence, Stress
Keywords: bulking agent; emivulvectomy; radical vulvectomy; TVT; urinary incontinence; vulvar cancer
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Vulvar Neoplasms | interventions — Suburethral Slings

ARMS (2):
- Tension free vaginal tape (Active Comparator)
  Interventions: Procedure: Tension free vaginal tape
- Bulking agent injection (Experimental)
  Interventions: Procedure: Bulking agent injection

INTERVENTIONS:
Procedure: Tension free vaginal tape — Small incision sites in the vagina and suprapubically. Bilateral retropubic insertion of the sling by means of needles
  Arms: Tension free vaginal tape
Procedure: Bulking agent injection — Three Periurethral injections of Bulkamid ® (Ethicon,Somerville, NJ, USA)
  Arms: Bulking agent injection

SUMMARY:
The surgical treatment of vulvar cancer is characterized by a radical approach as standard, often associated to an important rate of functional complications. This surgery often includes the partial excision of urethra, resulting in a reduction of urethral closure pressure. The radiotherapy-induced fibrosis in addiction leads to a reduction of urethral mobility. As consequence women treated for vulvar cancer may develop urinary incontinence. The incidence of this complication has been differently reported, but seems to reach the 100%. Poor data are available regarding the treatment of post vulvectomy urinary incontinence and no clear indication may be given at regards.

Based on these considerations the aim of this trial will be to compare tension free vaginal tape and bulking agent injection in women with urinary stress incontinence developed after radical surgery for vulvar cancer.

DETAILED DESCRIPTION:
Women with urinary stress incontinence developed after radical vulvectomy will be enrolled and randomized in two groups (arm 1 and arm 2). Patients of group 1 will be treated with the tension free vaginal tape, whereas in patients of arm 2 will be used the bulking agent injection.

All eligible patients will undergo baseline assessment consisting of anthropometric, clinical, and urodynamic evaluations. During the study, the surgical outcomes, the clinical subjective and objective efficacy data, and the adverse experiences will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Stress urinary incontinence by self report, examination and test
* History of radical vulvectomy

Exclusion Criteria:

* Systemic disease and/or drugs known to affect bladder function
* Current chemotherapy or radiation therapy
* Detrusor instability

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cure rate | 12 months

SECONDARY OUTCOMES:
Intra-operative complication rate | 1 day
Postoperative complication rate | 12 months
Recurrence rate | 12 months
Second surgery for stress urinary incontinence (SUI) | 12 months
Quality of life | 12 months
Satisfaction | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pugliese Hospital, Catanzaro, Italy